CLINICAL TRIAL: NCT01981642
Title: Nicht-invasive Diagnostik in Patienten Mit Herzunterstützungssystemen
Brief Title: Noninvasive Diagnostics in Left Ventricular Assist Device Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Austrian Science Fund (FWF) (Other)
Responsible Party: Principal Investigator, Francesco Moscato, Assoc. Prof. Dipl.-Ing. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MUW_EK-243/2011; KLI357 (Other Grant/Funding Number: Austrian Science Fund (FWF))
Record Dates: First submitted 2013-10-29; First posted 2013-11-11 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure; Artificial Heart Device User
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with a LVAD implanted. (Experimental): Recording of LVAD data during routine visits and daily life. Recording of daily activity using wristwatch accelerometers.
  Interventions: Other: Recording of LVAD data during routine visits and daily life.; Other: Recording of daily activity using wristwatch accelerometers.

INTERVENTIONS:
Other: Recording of LVAD data during routine visits and daily life. — Noninvasive diagnostic intervention.
Other: Recording of daily activity using wristwatch accelerometers. — Noninvasive diagnostic intervention.

SUMMARY:
* Study Purpose: The purpose of this study is to evaluate the sensitivity/specificity of noninvasive diagnostic methods for the cardiac function that are based on data available from the Left Ventricular Assist Device (LVAD). These diagnostic methods will be compared to standard clinical diagnostic procedures both at rest and during exercise.
* Study Design: The study is a prospective interventional cohort study.
* Patient cohort: Thirty heart failure patients who had or are about to have a LVAD implanted.
* Data Collection: The acquisition of LVAD data (motor current and speed) and wristwatch accelerometry data concurrently to the documentation of routine clinical examinations, such as cardiac ultrasound, electrocardiography (ECG), cardiac catheterization, and exercise tests, will be performed.

DETAILED DESCRIPTION:
* Background: In recent years Left Ventricular Assist Devices (LVADs) have become the devices of choice to treat patients with advanced heart failure. Proper evaluation of the cardiovascular function under LVAD support is of key importance especially for the preservation of the assisted cardiac function or for the evaluation of an eventual cardiac recovery. Cardiac echocardiography, electrocardiography and catheterization, as well as exercise testing are the standard clinical methods for the evaluation of the cardiovascular function during LVAD support. All these methods require however time-consuming procedures, and are therefore unacceptably cumbersome for frequent monitoring. On the other hand, a frequent and effective noninvasive evaluation of the cardiac status provided by the LVAD itself would have a remarkable impact on LVAD patients and their therapy. Previously developed methods to assess the cardiovascular status from data available from the LVAD (see references given) will be now investigated in a prospective clinical study.
* Purpose: The main purpose of this study is evaluate the sensitivity/specificity of LVAD based diagnostics when compared to standard clinical diagnostic procedures both at rest and during exercise. Secondarily, the physical activity of patients will be evaluated following LVAD implantation.
* Methods: Seventy-five heart failure patients who had or are about to have a LVAD implanted will be enrolled in this study. In these patients, the LVAD data (motor current and speed) will be recorded concurrently to the routine clinical examinations and during daily life. The routine clinical examinations typically consist of a subset of the following procedures: cardiac ultrasound, cardiac catheterization, 24h ECG measurement, exercise tests (6-minute walk test and spiroergometry). Parameters from the LVAD data that reflect contractile and relaxation properties as well as and aortic valve opening will be compared to echocardiography. Parameters from the LVAD data that reflect cardiac rhythms will be compared to ECG measurements. Both cardiac hemodynamics and rhythms during exercise tests will be assessed using the developed methods based on LVAD data. Finally, wristwatch accelerometers will be used for a quantification and evaluation of patient daily life activity. This measurements will be compared to 6-minute walk test and spiroergometry data as well as with the diagnostics methods based on the LVAD data.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained from the subject prior to participation;
* At least 18 years of age and maximum 70 years old;
* Subjects who received or are about to receive an LVAD.

Exclusion Criteria:

* Coagulation system disorders;
* Pregnant or breast-feeding women;
* Patients with bi-ventricular assist devices.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity/specificity of LVAD-based methods to monitor the cardiovascular function when compared to routine clinical diagnostics. | Participants will be followed for the duration of LVAD implant, an expected average of 2 years.

SECONDARY OUTCOMES:
Documentation of daily life activities as measured using wristwatch accelerometers and routine clinical exercise tests. | Participants will be followed for the duration of LVAD implant, an expected average of 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Moscato, PhD, Principal Investigator — Medical University of Vienna; Daniel Zimpfer, MD, Principal Investigator — Medical University of Vienna; Heinrich Schima, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- General Hospital / Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Granegger M, Schima H, Zimpfer D, Moscato F. Assessment of aortic valve opening during rotary blood pump support using pump signals. Artif Organs. 2014 Apr;38(4):290-7. doi: 10.1111/aor.12167. Epub 2013 Sep 19. PMID 24102321
- [Background] Moscato F, Granegger M, Edelmayer M, Zimpfer D, Schima H. Continuous monitoring of cardiac rhythms in left ventricular assist device patients. Artif Organs. 2014 Mar;38(3):191-8. doi: 10.1111/aor.12141. Epub 2013 Aug 1. PMID 23902542
- [Background] Granegger M, Moscato F, Casas F, Wieselthaler G, Schima H. Development of a pump flow estimator for rotary blood pumps to enhance monitoring of ventricular function. Artif Organs. 2012 Aug;36(8):691-9. doi: 10.1111/j.1525-1594.2012.01503.x. PMID 22882439
- [Background] Moscato F, Granegger M, Naiyanetr P, Wieselthaler G, Schima H. Evaluation of left ventricular relaxation in rotary blood pump recipients using the pump flow waveform: a simulation study. Artif Organs. 2012 May;36(5):470-8. doi: 10.1111/j.1525-1594.2011.01392.x. Epub 2011 Dec 16. PMID 22171892
- [Background] Naiyanetr P, Moscato F, Vollkron M, Zimpfer D, Wieselthaler G, Schima H. Continuous assessment of cardiac function during rotary blood pump support: a contractility index derived from pump flow. J Heart Lung Transplant. 2010 Jan;29(1):37-44. doi: 10.1016/j.healun.2009.05.032. Epub 2009 Sep 26. PMID 19782591
- [Background] Vollkron M, Schima H, Huber L, Benkowski R, Morello G, Wieselthaler G. Advanced suction detection for an axial flow pump. Artif Organs. 2006 Sep;30(9):665-70. doi: 10.1111/j.1525-1594.2006.00282.x. PMID 16934094
- [Derived] Berger L, Haberbusch M, Gross C, Moscato F. Enhancing Heart Failure Care: Deep Learning-Based Activity Classification in Left Ventricular Assist Device Patients. ASAIO J. 2025 Jan 1;71(1):52-60. doi: 10.1097/MAT.0000000000002299. Epub 2024 Sep 4. PMID 39231213